CLINICAL TRIAL: NCT06706947
Title: Exploration of the Efficacy and Mechanisms of Lymphaticovenous Anastomosis in the Treatment of Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luo Xinxin (Other)
Collaborators: Shenzhen Bao'an People's Hospital (Unknown); Shenzhen Kangning Hospital (Other)
Responsible Party: Sponsor-Investigator, Luo Xinxin, Director, Zhongshan Third People's Hospital
Organization: Zhongshan Third People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSYLL-KY-20241002
Record Dates: First submitted 2024-11-06; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer's Disease (AD)
Keywords: Lymphaticovenous Anastomosis; cognitive function; therapeutic efficacy; Mechanism; Alzheimer's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lymphaticovenous Anastomosis (Experimental)
  Interventions: Procedure: Lymphaticovenous Anastomosis

INTERVENTIONS:
Procedure: Lymphaticovenous Anastomosis — Lymphaticovenous Anastomosis (LVA) is an emerging super-microsurgical procedure pioneered by Professor Xie Qingping and his team, a group of Chinese microsurgery experts. This technique has been published in the official journal of the American Society of Plastic Surgeons (ASPS), confirming its effectiveness in improving the "drainage" function of the brain and reducing lymphatic pressure in deep brain tissues. By establishing an anastomosis between lymphatic vessels and veins in the neck, the surgery enhances the drainage of cerebrospinal fluid, alleviating the accumulation of toxins and waste within the brain, thereby easing the symptoms of Alzheimer's disease. Due to its significant contribution to the field of microsurgery, this innovative surgery has been selected as one of the "Top Seven Advances in Microsurgery for 2022."
  Other Names: LVA

SUMMARY:
The aim of this clinical trial is to determine whether Lymphaticovenous Anastomosis can treat Alzheimer's disease，in AD patients aged 18-80.he main questions it aims to answer are:

1. Can Lymphaticovenous Anastomosis improve cognitive function, daily living ability, mood, or sleep status in patients with Alzheimer's dementia, demonstrating good therapeutic efficacy?
2. Does deep Lymphaticovenous Anastomosis lead to changes in peripheral blood biomarker levels, neuroinflammatory responses, and neuroimaging in patients with Alzheimer's dementia?

ELIGIBILITY:
Inclusion Criteria:

1. At least two deputy chief physicians or above, diagnosed with Alzheimer's dementia according to the DSM-5 diagnostic criteria;
2. Age between 18-80 years old;
3. The course of the disease is at least 1 year;
4. MMSE score ≤ 24 points; MoCA score < 26
5. Brain MRI shows hippocampal atrophy;
6. Patients and their families agree to participate in this project for surgical treatment and sign an informed consent form.

Exclusion Criteria:

1. Individuals with contraindications for Lymphaticovenous Anastomosis; those allergic to anesthetics and contrast agents (indocyanine green);
2. Those unable to cooperate with cranial magnetic resonance imaging and scale testing;
3. Patients simultaneously suffering from schizophrenia, depression, bipolar disorder;
4. Patients with severe somatic diseases (such as cardiovascular, liver, kidney, gastrointestinal, etc.), infectious diseases, and immune system disorders;
5. Individuals with serious neurological diseases (such as epilepsy, cerebrovascular diseases, etc.), other types of dementia, mental retardation;
6. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination(MMSE) | half a year

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Third People's Hospital, Shenzhen, China

REFERENCES:
- [Background] Waldemar G, Phung KT, Burns A, Georges J, Hansen FR, Iliffe S, Marking C, Rikkert MO, Selmes J, Stoppe G, Sartorius N. Access to diagnostic evaluation and treatment for dementia in Europe. Int J Geriatr Psychiatry. 2007 Jan;22(1):47-54. doi: 10.1002/gps.1652. PMID 17044135
- [Background] Da Mesquita S, Louveau A, Vaccari A, Smirnov I, Cornelison RC, Kingsmore KM, Contarino C, Onengut-Gumuscu S, Farber E, Raper D, Viar KE, Powell RD, Baker W, Dabhi N, Bai R, Cao R, Hu S, Rich SS, Munson JM, Lopes MB, Overall CC, Acton ST, Kipnis J. Functional aspects of meningeal lymphatics in ageing and Alzheimer's disease. Nature. 2018 Aug;560(7717):185-191. doi: 10.1038/s41586-018-0368-8. Epub 2018 Jul 25. PMID 30046111
- [Background] Aspelund A, Antila S, Proulx ST, Karlsen TV, Karaman S, Detmar M, Wiig H, Alitalo K. A dural lymphatic vascular system that drains brain interstitial fluid and macromolecules. J Exp Med. 2015 Jun 29;212(7):991-9. doi: 10.1084/jem.20142290. Epub 2015 Jun 15. PMID 26077718
- [Background] Louveau A, Smirnov I, Keyes TJ, Eccles JD, Rouhani SJ, Peske JD, Derecki NC, Castle D, Mandell JW, Lee KS, Harris TH, Kipnis J. Structural and functional features of central nervous system lymphatic vessels. Nature. 2015 Jul 16;523(7560):337-41. doi: 10.1038/nature14432. Epub 2015 Jun 1. PMID 26030524
- [Background] Olate-Briones A, Escalona E, Salazar C, Herrada MJ, Liu C, Herrada AA, Escobedo N. The meningeal lymphatic vasculature in neuroinflammation. FASEB J. 2022 May;36(5):e22276. doi: 10.1096/fj.202101574RR. PMID 35344212
- [Background] Busch N, O'Reilly L, Louveau A. Meningeal Lymphatic vasculature in health and disease. Curr Opin Hematol. 2022 May 1;29(3):151-155. doi: 10.1097/MOH.0000000000000711. Epub 2022 Feb 18. PMID 35441600
- [Background] Alitalo K. The lymphatic vasculature in disease. Nat Med. 2011 Nov 7;17(11):1371-80. doi: 10.1038/nm.2545. PMID 22064427
- [Background] Iliff JJ, Wang M, Liao Y, Plogg BA, Peng W, Gundersen GA, Benveniste H, Vates GE, Deane R, Goldman SA, Nagelhus EA, Nedergaard M. A paravascular pathway facilitates CSF flow through the brain parenchyma and the clearance of interstitial solutes, including amyloid beta. Sci Transl Med. 2012 Aug 15;4(147):147ra111. doi: 10.1126/scitranslmed.3003748. PMID 22896675
- [Background] Zhang B, Gaiteri C, Bodea LG, Wang Z, McElwee J, Podtelezhnikov AA, Zhang C, Xie T, Tran L, Dobrin R, Fluder E, Clurman B, Melquist S, Narayanan M, Suver C, Shah H, Mahajan M, Gillis T, Mysore J, MacDonald ME, Lamb JR, Bennett DA, Molony C, Stone DJ, Gudnason V, Myers AJ, Schadt EE, Neumann H, Zhu J, Emilsson V. Integrated systems approach identifies genetic nodes and networks in late-onset Alzheimer's disease. Cell. 2013 Apr 25;153(3):707-20. doi: 10.1016/j.cell.2013.03.030. PMID 23622250
- [Background] Bai Y, Ma X. Chlorzoxazone exhibits neuroprotection against Alzheimer's disease by attenuating neuroinflammation and neurodegeneration in vitro and in vivo. Int Immunopharmacol. 2020 Nov;88:106790. doi: 10.1016/j.intimp.2020.106790. Epub 2020 Aug 11. PMID 32795892
- [Background] Park J, Wetzel I, Marriott I, Dreau D, D'Avanzo C, Kim DY, Tanzi RE, Cho H. A 3D human triculture system modeling neurodegeneration and neuroinflammation in Alzheimer's disease. Nat Neurosci. 2018 Jul;21(7):941-951. doi: 10.1038/s41593-018-0175-4. Epub 2018 Jun 27. PMID 29950669
- [Background] Mummery CJ, Borjesson-Hanson A, Blackburn DJ, Vijverberg EGB, De Deyn PP, Ducharme S, Jonsson M, Schneider A, Rinne JO, Ludolph AC, Bodenschatz R, Kordasiewicz H, Swayze EE, Fitzsimmons B, Mignon L, Moore KM, Yun C, Baumann T, Li D, Norris DA, Crean R, Graham DL, Huang E, Ratti E, Bennett CF, Junge C, Lane RM. Tau-targeting antisense oligonucleotide MAPTRx in mild Alzheimer's disease: a phase 1b, randomized, placebo-controlled trial. Nat Med. 2023 Jun;29(6):1437-1447. doi: 10.1038/s41591-023-02326-3. Epub 2023 Apr 24. PMID 37095250
- [Background] Mintun MA, Lo AC, Duggan Evans C, Wessels AM, Ardayfio PA, Andersen SW, Shcherbinin S, Sparks J, Sims JR, Brys M, Apostolova LG, Salloway SP, Skovronsky DM. Donanemab in Early Alzheimer's Disease. N Engl J Med. 2021 May 6;384(18):1691-1704. doi: 10.1056/NEJMoa2100708. Epub 2021 Mar 13. PMID 33720637
- [Background] Panza F, Lozupone M, Seripa D, Imbimbo BP. Amyloid-beta immunotherapy for alzheimer disease: Is it now a long shot? Ann Neurol. 2019 Mar;85(3):303-315. doi: 10.1002/ana.25410. Epub 2019 Jan 28. PMID 30635926
- [Background] Zhang ZX, Zahner GE, Roman GC, Liu XH, Wu CB, Hong Z, Hong X, Tang MN, Zhou B, Qu QM, Zhang XJ, Li H. Socio-demographic variation of dementia subtypes in china: Methodology and results of a prevalence study in Beijing, Chengdu, Shanghai, and Xian. Neuroepidemiology. 2006;27(4):177-87. doi: 10.1159/000096131. Epub 2006 Oct 11. PMID 17035714
- [Background] Huang Y, Wang Y, Wang H, Liu Z, Yu X, Yan J, Yu Y, Kou C, Xu X, Lu J, Wang Z, He S, Xu Y, He Y, Li T, Guo W, Tian H, Xu G, Xu X, Ma Y, Wang L, Wang L, Yan Y, Wang B, Xiao S, Zhou L, Li L, Tan L, Zhang T, Ma C, Li Q, Ding H, Geng H, Jia F, Shi J, Wang S, Zhang N, Du X, Du X, Wu Y. Prevalence of mental disorders in China: a cross-sectional epidemiological study. Lancet Psychiatry. 2019 Mar;6(3):211-224. doi: 10.1016/S2215-0366(18)30511-X. Epub 2019 Feb 18. PMID 30792114
- [Background] Alzheimer's Association. 2016 Alzheimer's disease facts and figures. Alzheimers Dement. 2016 Apr;12(4):459-509. doi: 10.1016/j.jalz.2016.03.001. PMID 27570871
- [Background] Li D, Zhang DJ, Shao JJ, Qi XD, Tian L. A meta-analysis of the prevalence of depressive symptoms in Chinese older adults. Arch Gerontol Geriatr. 2014 Jan-Feb;58(1):1-9. doi: 10.1016/j.archger.2013.07.016. Epub 2013 Aug 13. PMID 24001674
- [Background] Alzheimer's Association. 2014 Alzheimer's disease facts and figures. Alzheimers Dement. 2014 Mar;10(2):e47-92. doi: 10.1016/j.jalz.2014.02.001. PMID 24818261
- [Background] Hugo J, Ganguli M. Dementia and cognitive impairment: epidemiology, diagnosis, and treatment. Clin Geriatr Med. 2014 Aug;30(3):421-42. doi: 10.1016/j.cger.2014.04.001. Epub 2014 Jun 12. PMID 25037289